CLINICAL TRIAL: NCT01332097
Title: An Exploratory, Randomized, Double-blind, Placebo Controlled, Multi-center Study to Assess the Efficacy, Safety and Tolerability of a Single and a Repeated Dose of Oral BCT197 in Patients With an Acute COPD Exacerbation
Brief Title: Safety & Efficacy of BCT197A2201 in COPD Patients Presenting With an Exacerbation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBCT197A2201; 2010-021723-27 (EudraCT Number)
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Exacerbation; Pulmonary Inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): Single 75mg oral dose of BCT197 capsules + single oral dose of prednisone placebo capsules
  Interventions: Drug: BCT197; Drug: Prednisone placebo
- Treatment B/G/E/I (Placebo Comparator): Matching placebo comparator arm
  Interventions: Drug: Prednisone placebo; Drug: BCT197 placebo
- Treatment C (Active Comparator): Single oral dose of BCT 197 placebo capsules + single oral dose of 40mg prednisone capsules
  Interventions: Drug: BCT197 placebo; Drug: Prednisone
- Treatment D (Experimental): Single oral dose of 20mg dose of BCT197 capsules
  Interventions: Drug: BCT197
- Treatment F (Experimental): Single oral dose of 20 mg dose of BCT197 capsules on Day 1 and Day 6
  Interventions: Drug: BCT197
- Treatment H (Experimental): Single oral dose of 75mg dose of BCT197 capsules on Day 1 and Day 6
  Interventions: Drug: BCT197

INTERVENTIONS:
Drug: BCT197
  Arms: Treatment A; Treatment D; Treatment F; Treatment H
Drug: Prednisone placebo — capsules
  Arms: Treatment A; Treatment B/G/E/I
Drug: BCT197 placebo — capsules
  Arms: Treatment B/G/E/I; Treatment C
Drug: Prednisone — capsules
  Arms: Treatment C

SUMMARY:
This study will assess preliminary parameters of safety and efficacy of a single dose of BCT197 in patients with a Chronic Obstructive Pulmonary Disease (COPD) exacerbation.

DETAILED DESCRIPTION:
This was an exploratory, double-blind, randomized, placebo-controlled, multicenter, adaptive parallel-group design study in four parts in patients with acute COPD exacerbation. In Part I, patients were randomized to receive either a single dose of 75mg BCT197, placebo or 40 mg oral prednisone in the ratio of 1:1:1. In Part II patients were randomized to receive either a single dose of 20 mg BCT197 or placebo in the ratio of 5:1. Patients in Parts I and II received their single dose on Day 1 of the study. In Parts III and IV patients were randomized to receive either BCT197 or placebo in a ratio of 5:1 at a dose of 20mg (Part III) or 75 mg (Part IV) with patients receiving a single dose on both Day 1 and Day 6 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD (Stage II to IV) with a COPD exacerbation.
* Smoking history of 10 pack years.
* Females must not be of child-bearing potential.

Exclusion Criteria:

* Use of steroids in the last 30 days or calcium channel blockers in the last 48 hours.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Parkin, PhD FRCP, Study Director — Mereo BioPharma
Locations (5):
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
- Novartis Investigative Site, Bucharest, Romania
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strambu IR, Kobalava ZD, Magnusson BP, MacKinnon A, Parkin JM. Phase II Study of Single/Repeated Doses of Acumapimod (BCT197) to Treat Acute Exacerbations of COPD. COPD. 2019 Dec;16(5-6):344-353. doi: 10.1080/15412555.2019.1682535. Epub 2019 Nov 4. PMID 31682162

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: Single 75mg oral dose of BCT197 capsules + single oral dose of prednisone placebo capsules
  BCT197
  Prednisone placebo: capsules
- Treatment C: Single oral dose of BCT 197 placebo capsules + single oral dose of 40mg prednisone capsules
  Prednisone placebo: capsules
  BCT197 placebo: capsules
- Treatment D: Single oral dose of 20mg dose of BCT197 capsules
  BCT197
- Treatment F: Single oral dose of 20 mg dose of BCT197 capsules on Day 1 and Day 6
  BCT197
- Treatment H: Single oral dose of 75mg dose of BCT197 capsules on Day 1 and Day 6
  BCT197
- Treatment B,E,G I: Matching placebo group Treatment B - Single oral dose of BCT placebo Treatment E - Single oral dose of BCT197 placebo and prednisone placebo Treatment G - Single oral dose of BCT197 placebo and Treatment I - Single oral dose of BCT197 placebo
Period: Overall Study
Arm/Group | Treatment A | Treatment C | Treatment D | Treatment F | Treatment H | Treatment B,E,G I
Started | 31 | 30 | 25 | 27 | 25 | 45
Completed | 30 | 26 | 23 | 24 | 22 | 44
Not Completed | 1 | 4 | 2 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment B, E,G & I: Matched placebo arms
  BCT197 placebo: capsules
  Prednisone placebo: capsules
- Treatment C: Single oral dose of BCT197 placebo capsules + single oral dose of 40mg prednisone capsules
  Prednisone: capsules
  BCT197 placebo: capsules
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B, E,G & I | Treatment C | Treatment D | Treatment F | Treatment H | Total
Number analyzed (Participants) | 31 | 45 | 30 | 25 | 27 | 25 | 183
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (8.6) | 61 (6.6) | 63 (8.0) | 62 (8.7) | 61 (9.1) | 64 (6.7) | 62 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 4 | 4 | 4 | 4 | 37
  Male | 23 | 32 | 26 | 21 | 23 | 21 | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 31 | 45 | 30 | 25 | 27 | 25 | 183
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1 From Baseline to Day 5 or Baseline to Day 10 Measure: FEV1 Change in Forced Expiry Volume in 1 Second
Description: Change in FEV1 from baseline to Day 5 or baseline to Day 10 measured in mL
  Measure: FEV1
  Change in Forced Expiry Volume in 1 second
Time Frame: Day 5, Day 10
Population: The PD analysis set included all participants without major protocol deviations that impacted efficacy/pharmacodynamic data. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and "Number analyzed" is the number of participants evaluated at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Groups:
- Treatment B, E, G & I: Matched Placebo arms
  BCT197 placebo: capsules
  Prednisone placebo: capsules
- Treatment C: Single oral dose of BCT197 placebo capsules + single oral dose of 40mg prednisone capsules
  Prednisone
  BCT197 placebo: capsules
Arm/Group | Treatment A | Treatment B, E, G & I | Treatment C | Treatment D | Treatment F | Treatment H
Number analyzed (Participants) | 30 | 45 | 30 | 25 | 26 | 25
mL
  Day 5 | 155.1 [80.8 to 229.3] | 100.8 [40.0 to 161.7] | 48.9 [-25.6 to 123.3] | 106.3 [24.7 to 187.9] | 134.4 [54.6 to 214.1] | 200.6 [119.0 to 282.3]
  Day 10: number analyzed (Participants) | 14 | 24 | 15 | 7 | 26 | 25
  Day 10 | 164.6 [51.0 to 278.3] | 126.9 [37.0 to 216.8] | 54.9 [-56.8 to 166.7] | 54.6 [-88.8 to 198.0] | 109.0 [5.6 to 212.5] | 250.5 [144.5 to 356.4]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B, E, G & I; LS Mean difference: Treatment A vs. Treatment B, E, G & I (placebo) Day 5; Test type: Superiority; Least squares mean difference = 54.2, 95% CI 2-sided [-41.7 to 150.1]
Statistical Analysis 2: Comparison: Treatment B, E, G & I vs Treatment C; LS Mean difference: Treatment C vs. Treatment B, E, G & I (placebo) Day 5; Test type: Superiority; Least squares mean difference = -52.0, 95% CI 2-sided [-148.5 to 44.5]
Statistical Analysis 3: Comparison: Treatment B, E, G & I vs Treatment D; LS Mean difference: Treatment D vs. Treatment B, E, G & I (placebo) Day 5; Test type: Superiority; Least squares mean difference = 5.5, 95% CI 2-sided [-96.0 to 106.9]
Statistical Analysis 4: Comparison: Treatment B, E, G & I vs Treatment F; LS Mean difference: Treatment F vs. Treatment B, E, G & I (placebo) Day 5; Test type: Superiority; Least squares mean difference = 33.5, 95% CI 2-sided [-66.8 to 133.9]
Statistical Analysis 5: Comparison: Treatment B, E, G & I vs Treatment H; LS Mean difference: Treatment H vs. Treatment B, E, G & I (placebo) Day 5; Test type: Superiority; Least squares mean difference = 99.8, 95% CI 2-sided [-2.4 to 202.0]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B, E, G & I; LS Mean difference: Treatment A vs. Treatment B, E, G & I (placebo) Day 10; Test type: Superiority; Least squares mean difference = 37.8, 95% CI 2-sided [-107.1 to 182.6]
Statistical Analysis 7: Comparison: Treatment B, E, G & I vs Treatment C; LS Mean difference: Treatment C vs. Treatment B, E, G & I (placebo) Day 10; Test type: Superiority; Least squares mean difference = -72.0, 95% CI 2-sided [-215.7 to 71.8]
Statistical Analysis 8: Comparison: Treatment B, E, G & I vs Treatment D; LS Mean difference: Treatment D vs. Treatment B, E, G & I (placebo) Day 10; Test type: Superiority; Least squares mean difference = -72.3, 95% CI 2-sided [-241.5 to 96.9]
Statistical Analysis 9: Comparison: Treatment B, E, G & I vs Treatment F; LS Mean difference: Treatment F vs. Treatment B, E, G & I (placebo) Day 10; Test type: Superiority; Least squares mean difference = -17.9, 95% CI 2-sided [-154.9 to 119.2]
Statistical Analysis 10: Comparison: Treatment B, E, G & I vs Treatment H; LS Mean difference: Treatment H vs. Treatment B, E, G & I (placebo) Day 10; Test type: Superiority; Least squares mean difference = 123.6, 95% CI 2-sided [-15.8 to 263.0]

2. Secondary Outcome: Rolling Average Improvement From Day 1 to Day 29 Using the EXACT-PRO 14 Point Patient Reported Outcome Measure: EXACT-PRO
Description: EXAcerbations of Chronic pulmonary disease tool patient reported outcome (EXACT-PRO) Rolling Average Improvement from Day 1 to Day 29. EXACT-PRO is a 14 point patient reported daily diary used to quantify and measure exacerbations of chronic obstructive pulmonary disease (COPD). Minimum score is 0 and Maximum score is 14 (higher scores indicate worsening indicative of an exacerbation). Reported value is LS mean improvement from at Day 29 compared to D1 of the study.
Time Frame: Up to Day 29
Population: The PD analysis set included all participants without major protocol deviations that impacted efficacy/pharmacodynamic data. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment A | Treatment B, E, G & I | Treatment C | Treatment D | Treatment F | Treatment H
Number analyzed (Participants) | 25 | 41 | 26 | 23 | 24 | 24
score on a scale | 5.72 [0.55 to 10.90] | 8.89 [4.74 to 13.05] | 5.19 [0.02 to 10.36] | 5.83 [-0.35 to 12.01] | 7.89 [2.58 to 13.20] | 8.35 [2.59 to 14.11]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Treatment B, E, G & I: Matching placebo
  Single oral dose of BCT197 placebo capsules + single oral dose of prednisone placebo capsules
  Prednisone placebo: capsules
  BCT197 placebo: capsules
Arm/Group | Treatment A | Treatment B, E, G & I | Treatment C | Treatment D | Treatment F | Treatment H
All-Cause Mortality (participants affected / at risk) | 1/31 | 0/45 | 2/30 | 1/25 | 1/27 | 1/25
Serious Adverse Events (participants affected / at risk) | 2/31 | 4/45 | 5/30 | 2/25 | 3/27 | 3/25
Other Adverse Events (participants affected / at risk) | 5/31 | 20/45 | 16/30 | 13/25 | 14/27 | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=31) | Treatment B, E, G & I (N=45) | Treatment C (N=30) | Treatment D (N=25) | Treatment F (N=27) | Treatment H (N=25)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 3 (4) | 1 (1) | 2 (3) | 3 (4) — COPD Exacerbation
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Acute cardiac failure
Cerebral Edema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Brain odema
Decompensated Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Chronic respiratory failure
Attrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Attrial Flutter
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Sudden cardiac death
Stoke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Cerebrovascular accident
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=31) | Treatment B, E, G & I (N=45) | Treatment C (N=30) | Treatment D (N=25) | Treatment F (N=27) | Treatment H (N=25)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Occult blood (Investigations) | 3 (3) | 3 (3) | 3 (3) | 5 (5) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (12) | 5 (5) | 4 (4) | 5 (5) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs must seek written permission from the sponsor before publication of any trial results.